CLINICAL TRIAL: NCT03466554
Title: Hyperbaric Oxygen Therapy for Adult Onset Post Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shay Efrati, head of segol center, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 199-17
Record Dates: First submitted 2018-03-04; First posted 2018-03-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Ptsd
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric oxygen therapy (HBOT) active treatment (Experimental): 60 daily HBOT sessions will be administrated 5 days per week. Comprise of 90 minutes exposure to 100% oxygen at 2 ATA, with 5-minute air breaks every 20 minutes.
  Interventions: Device: Hyperbaric oxygen-90 minutes exposure to 100% oxygen at 2 ATA, with 5-minute air breaks every 20 minutes
- Control-follow up (No Intervention): The standard of care of psychological and mediational support .
  After 3 months of follow up, participants will be re-evaluated. The individuals in the control group will then be offered to receive the treatment and to be re-reevaluated after the treatment is over (3 months).

INTERVENTIONS:
Device: Hyperbaric oxygen-90 minutes exposure to 100% oxygen at 2 ATA, with 5-minute air breaks every 20 minutes — 60 daily HBOT sessions will be administrated 5 days per week. comprise of 90 minutes exposure to 100% oxygen at 2 ATA, with 5-minute air breaks every 20 minutes.
  Arms: hyperbaric oxygen therapy (HBOT) active treatment

SUMMARY:
Posttraumatic stress disorder (PTSD) is the long term effect of severely distressing traumatic event characterized by intrusive thoughts, nightmares, and avoidance. Brain imaging of PTSD patients demonstrate alterations in regional brain perfusion, with stunned, hypoperfused regions. Those brain-biological pathologies may be responsible for the limited success rate of currently available interventions.

During the last years data regarding Hyperbaric Oxygen Therapy (HBOT) induced neuroplasticity accumulated. A number of studies in traumatic brain injury, cerebrovascular attacks, and fibromyalgia have presented evidence of improved perfusion and recovery of metabolic brain tissues, accompanied by clinical improvement under HBOT even years after the acute insults.

Considerable evidence supports potential benefit of HBOT on PTSD, however, no clinical trial was done on this pure PTSD population. The aim of the proposed study is to examine hyperbaric oxygen therapy as a treatment for PTSD. Advanced brain imaging and functional analysis tools will be used to evaluate treatment's effect.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) has been described as "the complex somatic, cognitive, affective, and behavioral effects of psychological trauma". PTSD is triggered by a severe distressing traumatic event, in which an overwhelming amount of stress exceeds the ability of the individual to cope or integrate the emotions involved in the experience. The fact that a large portion of the affected population is previously healthy, young people who were thrown off their life course, contribute to the great motivation for research in this field. But unfortunately, the current available treatment improve some of the symptoms in only 32-66% of patients, and even after treatment, up to 60% still meet PTSD diagnosis.

In the last few years, there is growing knowledge regarding the neuro-biological changes that characterize PTSD. Brain imaging demonstrates alterations in regional brain perfusion, with stunning, hypoperfused regions. Those enduring brain-biological pathologies may explain the limited success rate of currently available interventions.

Accumulating studies presents evidence that hyperbaric oxygen therapy (HBOT) can induce neuroplasticity and recovery of metabolic injured brain tissues, even years after the acute insults. HBOT can initiate several brain-repair related mechanisms including brain angiogenesis; improve cerebral vascular flow enable regeneration of axonal white matter, stimulate axonal growth, promote blood-brain barrier integrity and reduce inflammatory reactions, as well as in brain edema.

The potential beneficial effects of HBOT were demonstrated in several clinical trials of traumatic brain injury(TBI)/post-concussion patients. Some of these trials, especially those in veterans, included patients who, in addition to post-concussion syndrome, had PTSD; as it is estimated that half of the soldiers with post-concussion syndrome due to mild TBI also meet the criteria of PTSD.

The aim of the proposed study is to evaluate the effect of HBOT on PTSD symptoms in adults with treatment resistant PTSD who were not exposed to TBI or blast injury. In addition to the clinical outcome, brain functionality and microstructure will also be evaluated by PET and DTI-MRI in order to shed additional light on the pathophysiology of PTSD and its response to treatment.

Study protocol:

Thirty male patients with adult onset PTSD, defined by DSM-V criteria, as a result of combat or a terror- related event, will be recruited to the study. Further criteria for study inclusion will be: age 25-60 years, 4-years or more from the traumatic event and failure to improve with at least one line of conventional treatment.

Study exclusion criteria will be: a history of traumatic brain injury or blast injury, epilepsy, a brain tumor; skull base fractures or neurosurgery, severe substance use disorders, a current manic episode, psychotic disorders or serious suicidal ideation at baseline; or major cognitive deficits; a history of HBOT for any reason prior to study enrollment; chest pathology incompatible with pressure changes (including active asthma); inner ear disease; the inability to perform an awake brain MRI test; and the inability to provide informed consent.

After recruitment, participants will be randomized to one of two study groups . A treatment group will proceed to a course of HBOT, while participants in the control group will continue with the current standard of care of psychiatric support and medications. After 3 months of follow up, participants of both groups will be re-evaluated. The individuals in the control group will then be offered to receive the treatment and to be re-reevaluated after the treatment is over (3 months). Further evaluation will be done at 6 and 12 month to evaluate long term effects of the treatment. During the study, all participant will continue with their current medications unless otherwise advise by their treating physician.

According to the HBOT protocol, 60 daily HBOT sessions will be administrated 5 days per week. Comprise of 90 minutes exposure to 100% oxygen at 2 ATA, with 5-minute air breaks every 20 minutes.

Study end points:

Primary end point PTSD symptoms, as assessed by the PTSD questionnaire

Secondary end points

1. Sleep disorders questionnaire: Medical Outcome Sleep Scale (MOS)
2. Quality of life and mood questionnaires: Patient global impression of change, SF-36, EQ-5D, SCL51
3. Diary for daily documentation of symptoms
4. Cognitive function- Cognitive function will be evaluated by the mainstreams Cognitive Health Assessment.
5. Brain imaging Brain imaging will include 2 types of imaging: perfusion magnetic resonance imaging (MRI) + diffusion tensor imaging (DTI), including resting state functional MRI and brain single photon emission computed tomography (PET-CT).

   5.1 Perfusion MRI+DTI and Resting state fMRI (rsfMRI) a method of functional brain imaging that can be used to evaluate regional interactions that occur when a participant is not performing an explicit task. This resting brain activity is observed by means of changes in blood flow in the brain, which creates what is referred to as a blood-oxygen-level dependent (BOLD) signal that can be measured using functional MRI (fMRI). +task 5.2 PET CT
6. Physiological evaluation of brain functionality using transcranial magnetic stimulation (TMS)-EEG examination:

This examination includes non-invasive safe brain monitoring and stimulation for the assessment of changes in brain functionality and connectivity. The procedure includes placement of EEG electrodes on an individual's head and measurement of the TMS-evoked electrophysiological response in the various brain regions. The examination takes about 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult onset PTSD, defined by DSM-V criteria, as a result of combat or a terror- related event.
* Age 25-60 years, 4-years or more from the traumatic event and failure to improve with at least one line of conventional treatment.

Exclusion Criteria:

* A history of traumatic brain injury, epilepsy, a brain tumor; skull base fractures or neurosurgery.
* Severe substance use disorders a current manic episode, psychotic disorders or serious suicidal ideation at baseline.
* Major cognitive deficits
* History of HBOT for any reason, prior to study enrollment.
* Chest pathology incompatible with pressure changes (including active asthma).
* Inner ear disease.
* The inability to perform an awake brain MRI test.
* Inability to provide informed consent

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms | at baseline and after 3 months
  Symptoms assessed by the PTSD questionnaire (0-80)

SECONDARY OUTCOMES:
Change in Sleep disorders questionnaire | at baseline and after 3 months
  Medical Outcome Sleep Scale (MOS) (0-100) higher values represent a better outcome
Change in Cognitive function | at baseline and after 3 months
  mainstreams Cognitive Health Assessment (values normalized for age and gender, with mean value of 100 and standard deviation of 15)
Change in Brain imaging | at baseline and after 3 months
  Brain imaging will include 2 types of imaging: perfusion magnetic resonance imaging (MRI) + diffusion tensor imaging (DTI), including resting state functional MRI and brain single photon emission computed tomography (PET-CT).
change in symptoms assessed by Diary for daily documentation of symptoms | at baseline and after 3 months
  VAS based mood score higher values represent a worse outcome
Change in Physiological evaluation of brain functionality | at baseline and after 3 months
  This examination includes non-invasive safe brain monitoring and stimulation for the assessment of changes in brain functionality and connectivity. The procedure includes placement of EEG electrodes on an individual's head and measurement of the TMS-evoked electrophysiological response in the various brain regions.

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No